CLINICAL TRIAL: NCT00800696
Title: Preventive Oral Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: this study was not initiated due to lack of funding
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Hilla Ben-Pazi, PI, Shaare Zedek Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 58/08
Record Dates: First submitted 2008-11-30; First posted 2008-12-02 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Fever; Respiratory Infection
Keywords: antibiotics; Hospitalization; oral care
MeSH Terms: conditions — Fever; Respiratory Tract Infections | interventions — Dental Care Team

ARMS (2):
- oral care (Experimental): intervention: The study group will have their teeth brushed three times a day by the nursing staff by using a suction connected toothbrush, daily examination of the oropharynx by the nursing staff, and use of chlorhexidine varnish or another suitable antibacterial agent in the oropharynx.
  Interventions: Procedure: oral care
- control (No Intervention): continue to receive oral care as performed today.

INTERVENTIONS:
Procedure: oral care — The study group will have their teeth brushed three times a day by the nursing staff by using a suction connected toothbrush, daily examination of the oropharynx by the nursing staff, and use of chlorhexidine varnish or another suitable antibacterial agent in the oropharynx
  Arms: oral care

SUMMARY:
The purpose of the investigators project is to examine if the investigators may affect a reduction in respiratory infections in a pediatric long term care facility by institution of a comprehensive oral care program. The investigators wish to base their project on work such as of Yoneyama et al 2002, which hypothesized and showed that "silent" aspiration of oropharyngeal contents is a causative factor in development of respiratory infection in elderly institutionalized clients. It was found that an advanced oral hygiene program greatly reduced the incidence of respiratory infection. Although no similar research projects were found to have involved children, the investigators hope that a similar program of oral care will allow the investigators to likewise reduce the incidence of respiratory infection among the pediatric clients in our facility.

The investigators propose to examine two groups of children which are fed by gastrostomy feedings only. One group will continue to receive oral care as performed today. The study group will have their teeth brushed three times a day by the nursing staff by using a suction connected toothbrush, daily examination of the oropharynx by the nursing staff, and use of chlorhexidine varnish or another suitable antibacterial agent in the oropharynx.

The investigators will retrospectively examine our records (a 12 month period) for febrile days, antibiotic use and hospitalization days due to respiratory causes. The investigators will then compare these to the febrile days, antibiotic use and hospitalizations to the 12 month period [post implementation of the oral care program.

The importance of this program is to examine whether by implementation of a relatively inexpensive and low-tech intervention may meaningfully reduce the morbidity and mortality due to respiratory infection among our clients (which from our experience is the main cause of morbidity and mortality in the investigators institution). The investigators expect that by reducing the incidence of respiratory disease among our clients that the investigators will greatly reduce suffering among the children and their families, improve their quality of life and ease the financial and organizational burdens as a result of caring for respiratory infections.

As was noted before, no prior research was found which studied the pediatric population in a long term care facilities. It is our belief that this project represents a unique research opportunity which may bring great benefit to the children and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Clients who receive gastrostomy feedings only
* ALEH Infirmary

Exclusion Criteria:

* Oral Feeding

Ages: 3 Months to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Hospitalization days per year | year

SECONDARY OUTCOMES:
Fever | year